CLINICAL TRIAL: NCT00538148
Title: A Multicenter, Multinational, Randomized, DB Controlled Study of the Efficacy & Safety of Oral Telithromycin 800 mg Once QD for 5 Days vs Azithromycin in the Treatment of Acute Exacerbation of Chronic Bronchitis in Adult Outpatients With COPD.
Brief Title: Telithromycin: in the Treatment of Acute Exacerbation of Chronic Bronchitis in Adult Outpatients With COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMR3647A_4014
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Bronchitis, Chronic
MeSH Terms: conditions — Bronchitis, Chronic | interventions — telithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Telithromycin

SUMMARY:
Non-inferiority efficacy of telithromycin versus azithromycin

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients, either sex, aged 45 years or older.
* Patients with a documented history of chronic bronchitis with a basal FEV1 <70% and >35% made in the previous 12 months and who had had at least one or more AEBC in the previous year and with FEV1/FVC <70% (lung function tests made in the previous 12 months).
* Patients with a clinical diagnosis of acute exacerbation of chronic bronchitis presumably due to bacterial infection based on all of the following signs and symptoms of AECB: increased sputum purulence, and at least 1 of the 2 following signs and symptoms (increased dyspnea, increased sputum volume).
* Patients with negative chest radiography (posterior/anterior and lateral views) to rule out a pneumonia within 48 hours before initiation of study medication or at the latest 24 hours after initiation of study medication (it was necessary to not include patients with pneumonia associated with AECB).
* Patients with sputum specimens collected at inclusion for gram stain and bacteriological culture.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2002-11; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Principal efficacy criterion: clinical outcome - Main secondary efficacy criteria: - Bacteriological response at TOC visit; - Time to relapse up to 6 months after inclusion. | At TOC visit (Day 17-Day 21).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi